CLINICAL TRIAL: NCT00003037
Title: Phase I/II Trial of the Combination of Docetaxel, Gemcitabine and Cisplatin (DGP) as Induction Chemotherapy in Patients With Stage III Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy as Induction Therapy in Treating Patients With Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 97-040; CDR0000065659 (Registry Identifier: PDQ (Physician Data Query)); NCI-G97-1285
Record Dates: First submitted 1999-11-01; First posted 2003-11-25 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel; Gemcitabine

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy with docetaxel, gemcitabine, and cisplatin as induction therapy in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) and schedule of docetaxel, gemcitabine, and cisplatin as induction chemotherapy in patients with Stage III non-small cell lung cancer (NSCLC) scheduled to undergo subsequent surgical resection or irradiation. II. Determine the major objective response rate of this combination therapy in these patients.

OUTLINE: This is a dose escalation study. Docetaxel in administered as a 1 hour IV infusion at week 1, 5, and 9. Gemcitabine is administered as a 30 minute IV infusion at weeks 1, 2, 3, 5, 6, 7, 9, 10, and 11. Cisplatin is administered as a 20 minute IV infusion at weeks 3, 7, and 11. In addition, G-CSF is administered subcutaneously on days 2 through 6 of each 28 day cycle following each dose of docetaxel. Three patients are entered at each dose level and must complete one cycle of therapy. If no patient experiences dose limiting toxicity (DLT), then 3 patients are treated at the next higher dose level. If 1 patient experiences DLT, then 3 more patients are treated at that same dose level. If 2 of 6 patients experience DLT, then that dose is declared the maximum tolerated dose (MTD). Once the MTD is determined, the Phase II portion of the study begins and additional patients are treated at the dose level just below the MTD. Patients who show complete or partial response, or no change, after chemotherapy, undergo surgical resection or radiotherapy to remove or reduce their tumor. Patients are assessed for disease progression and unacceptable toxicities every 4 weeks till end of treatment.

PROJECTED ACCRUAL: An estimated 40 patients will be accrued in this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed Stage III (T1-2 N2-3 M0, T3 N2 M0, or T4 N0-3 M0) non-small cell lung cancer Must be candidates for either a resection with curative intent or definitive thoracic irradiation following induction chemotherapy No malignant pericardial or pleural effusions or superior vena cava syndrome Must have measurable or evaluable indicator lesions

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 160,000/mm3 Hepatic: Bilirubin no greater than 1.0 mg/dL SGOT and/or SGPT no greater than 1.5 times the upper limit of normal Alkaline phosphatase no greater than 5 times the upper limit of normal Renal: Creatinine clearance at least 65 mL/min Cardiovascular: Must have stable heart rhythm No unstable angina No myocardial infarction within 6 months No clinical evidence of congestive heart failure Neurologic: Must have normal auditory function No symptoms of peripheral neuropathy Other: No prior malignancy except non-melanoma skin cancer or in situ carcinoma of the cervix Not pregnant Adequate contraception required of all fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiation therapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-04; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gomez, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States